CLINICAL TRIAL: NCT04080206
Title: An Open Label, Comparative Evaluation of the Adrenal Suppression Potential and Pharmacokinetic Properties of 188-0551 Spray Versus Reference Listed Drug (RLD) Applied Every 12 Hours for 2 Weeks in Subjects With Moderate to Severe Plaque Psoriasis
Brief Title: A Safety Study of 188-0551 Spray Versus Reference Listed Drug (RLD) in Adult Subjects With Plaque Psoriasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 188-0551-204
Record Dates: First submitted 2019-09-03; First posted 2019-09-06 (Actual); Last update posted 2021-05-10 (Actual); Status verified 2021-05

CONDITIONS: Plaque Psoriasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 188-0551 Spray (Experimental): Investigational Topical Spray Product
  Interventions: Drug: 188-0551 Spray
- Reference Listed Drug (RLD) (Active Comparator): FDA Approved Topical Cream
  Interventions: Drug: RLD

INTERVENTIONS:
Drug: 188-0551 Spray — Applied topically twice daily for two weeks
  Arms: 188-0551 Spray
Drug: RLD — Applied topically twice daily for two weeks
  Arms: Reference Listed Drug (RLD)

SUMMARY:
Adrenal suppression effects of corticosteroids are among the most important safety concerns for this group of products. This study is to determine and compare the adrenal suppression potential and the pharmacokinetic (PK) properties of 188-0551 Spray versus an FDA-approved drug (also known as a "Reference Listed Drug" [RLD]) under maximal use conditions when applied twice daily (approximately every 12 hours) in adult subjects with stable, moderate to severe, plaque psoriasis.

ELIGIBILITY:
Inclusion Criteria:

* Subject is a male or non-pregnant female and is at least 18 years of age at the time of informed consent.
* Subject has provided written informed consent.
* Subject has moderate or severe psoriasis involving a minimum of 20% Body Surface Area (BSA).
* Subject has an Investigator's Global Assessment (IGA) score of at least three (3 = moderate) at the Baseline Visit.

Exclusion Criteria:

* Subject is pregnant, lactating, or is planning to become pregnant during the study.
* Subject has spontaneously improving or rapidly deteriorating plaque psoriasis.
* Subject has a physical condition which, in the investigator's opinion, might impair evaluation of plaque psoriasis, adrenal axis function or which exposes the subject to an unacceptable risk by study participation.
* Subject has had prolonged exposure to natural or artificial sources of ultraviolet radiation.
* Subject is currently enrolled in an investigational drug or device study.
* Subject has clinically significant abnormal labs at Visit 1/Screening that precludes topical steroid use, in the opinion of the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2020-04-07 (Actual); Primary Completion 2021-01-20 (Actual); Study Completion 2021-01-20 (Actual)

PRIMARY OUTCOMES:
The proportion of subjects to exhibit adrenal suppression as measured by a cortrosyn stimulation test | Day 15
  A subject is considered to have adrenal suppression evidence if post stimulation lab draw result is ≤ 18 µg/dL (497 nmol/L).

CONTACTS AND LOCATIONS:
Locations (8):
- United States (3):
  - TI Site #13, Scottsdale, Arizona
  - TI Site #12, Thousand Oaks, California
  - TI Site #11, Miami, Florida
- Georgia (2):
  - TI Site #31, Batumi
  - TI Site #32, Tbilisi
- Ukraine (3):
  - TI Site #23, Lviv
  - TI Site #22, Rivne
  - TI Site #21, Zaporizhzhya

IPD SHARING:
Plan to Share IPD: No